CLINICAL TRIAL: NCT02400996
Title: A Single Centre Analysis of Clinical Characteristics and Treatment of Endocrine Pancreatic Tumours.
Brief Title: An Analysis of Presentation and Outcome Following Treatment of Pancreatic Endocrine Neoplasms
Status: Completed | Type: Observational
Sponsor: Medical College and Hospital Kolkata (Other)
Collaborators: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Md Tanveer Adil, Fellow, Sir Ganga Ram Hospital
Other Study IDs: SGRH-SGLT-MTA
Record Dates: First submitted 2015-03-23; First posted 2015-03-27 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatic Endocrine Neoplasms
Keywords: Endocrine Pancreas; Pancreatic Endocrine Neoplasm
MeSH Terms: conditions — Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic Endocrine Neoplasms: We did an observational analysis from a prospectively maintained database of patients who underwent pancreatic surgery for neoplasms of the pancreas at Sir Ganga Ram Hospital, New Delhi, India from 1995 to 2013 and using pathological reports and preoperative CT scan as gold standard, we identified 40 patients with PENs.

SUMMARY:
A single institutional study of Pancreatic Endocrine Neoplasms over 18 years.

DETAILED DESCRIPTION:
The investigators did an analysis from a prospectively maintained database of patients who underwent pancreatic resections or nonresective procedures for neoplasms of the pancreas at Sir Ganga Ram Hospital from 1995 to 2013 and using pathological reports and preoperative CT scan as the gold standard, the investigators identified 40 patients with PENs.

ELIGIBILITY:
Inclusion Criteria:

* Pathological reports and Prooperative CAT Scan showing Endocrine Pancreatic Tumours

Exclusion Criteria:

* Nonendocrine Pancreatic Tumours

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical files and electronic records were reviewed to collect information. Patients were categorized into functioning and nonfunctioning PENs based on their clinical behaviour, pathology reports and serum radioimmunoassay for offending hormones. Preoperative CT scans were used to characterize PENs and record neoplasm size and location in the pancreas. Review of operative notes was done for the type of surgery performed and peroperative findings recorded. Discharge summaries were used to study the surgical outcome in terms of duration of postoperative hospital stay and postoperative complications. Patients were followed up and any disease recurrence or disease related mortality was recorded. Evaluation of the pathology reports was done.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Md Tanveer Adil, Principal Investigator — Sir Ganga Ram Hospital, New Delhi; Raghavendra Nagaraja, Study Director — Sir Ganga Ram Hospital, New Delhi; Vibha Varma, Study Director — Sir Ganga Ram Hospital, New Delhi; Naimish Mehta, Study Director — Sir Ganga Ram Hospital, New Delhi; Vinay Kumaran, Study Director — Sir Ganga Ram Hospital, New Delhi; Samiran Nundy, Study Chair — Sir Ganga Ram Hospital, New Delhi

REFERENCES:
- [Background] Vortmeyer AO, Huang S, Lubensky I, Zhuang Z. Non-islet origin of pancreatic islet cell tumors. J Clin Endocrinol Metab. 2004 Apr;89(4):1934-8. doi: 10.1210/jc.2003-031575. PMID 15070966
- [Background] Halfdanarson TR, Rabe KG, Rubin J, Petersen GM. Pancreatic neuroendocrine tumors (PNETs): incidence, prognosis and recent trend toward improved survival. Ann Oncol. 2008 Oct;19(10):1727-33. doi: 10.1093/annonc/mdn351. Epub 2008 May 30. PMID 18515795
- [Result] Kazanjian KK, Reber HA, Hines OJ. Resection of pancreatic neuroendocrine tumors: results of 70 cases. Arch Surg. 2006 Aug;141(8):765-9; discussion 769-70. doi: 10.1001/archsurg.141.8.765. PMID 16924083
- [Result] Vagefi PA, Razo O, Deshpande V, McGrath DJ, Lauwers GY, Thayer SP, Warshaw AL, Fernandez-Del Castillo C. Evolving patterns in the detection and outcomes of pancreatic neuroendocrine neoplasms: the Massachusetts General Hospital experience from 1977 to 2005. Arch Surg. 2007 Apr;142(4):347-54. doi: 10.1001/archsurg.142.4.347. PMID 17438169
- [Result] Heitz PU, Komminoth P, Perrin A et al. Pancreatic endocrine tumors: Introduction. In: DeLellis DA, Lloyd RV, Heitz PU, et al., eds. Pathology and Genetics of Tumours of Endocrine Organs. WHO Classification of Tumours. Lyon, France: IARC Press, 2004: 177-82.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An analysis from a prospectively maintained database of patients was done who underwent pancreatic surgery for neoplasms of the pancreas at Sir Ganga Ram Hospital, New Delhi, India from 1995 to 2013 and using pathological reports and preoperative CT scan as gold standard, we identified 40 patients with PENs
Groups:
- Patients Operated for Pancreatic Endocrine Neoplasms: We did an observational analysis from a prospectively maintained database of patients who underwent pancreatic surgery for neoplasms of the pancreas at Sir Ganga Ram Hospital, New Delhi, India from 1995 to 2013 and using pathological reports and preoperative CT scan as gold standard, we identified 40 patients with PENs.
Period: Overall Study
Arm/Group | Patients Operated for Pancreatic Endocrine Neoplasms
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Operated for Pancreatic Endocrine Neoplasms
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (15.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 22
Region of Enrollment [Number; unit: participants]
  India | 40

OUTCOME MEASURES:

1. Primary Outcome: Nonfunctioning and Malignant Pancreatic Endocrine Neoplasms
Description: Of the 40 patients operated for Pancreatic Endocrine Neoplasms, using clinical criteria, histopathological analysis and preoperative imaging as gold standard, nonfunctioning and functioning tumours were identified. Similarly the number of benign and malignant lesions identified were recorded as per the WHO Classification of pancreatic endocrine tumours.
Time Frame: Each participant was followed up for a period of 5 years
Measure: Number; unit: participants
Arm/Group | Patients Operated for Pancreatic Endocrine Neoplasms
Number analyzed (Participants) | 40
participants
  Nonfunctioning Tumours | 28
  Functioning Tumours | 12
  Benign Tumours | 22
  Malignant Tumours | 18

ADVERSE EVENTS:
Time Frame: Complications were noted within the hospital admission. Postoperative mortality recorded as death within the same hospital admission or within 30 days of surgery. Follow up was done at 3 and 6 months and then at 6 monthly intervals for 5 years.
Description: The type of surgery performed, operative findings, postoperative hospital stay and complications were recorded. Postoperative mortality was recorded and followup done for disease recurrence or mortality.
Arm/Group | Pancreatic Endocrine Neoplasms
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 16/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pancreatic Endocrine Neoplasms (N=40)
Pancreatic fistula (Gastrointestinal disorders) | 6 (6) — A pancreatic fistula was defined as drainage of more than 30 mL of fluid per day with amylase levels at least 3 times the normal serum amylase levels from the sixth postoperative day
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pancreatic Endocrine Neoplasms (N=40)
Delayed Gastric Emptying (Gastrointestinal disorders) | 8 (8) — Delayed gastric emptying was defined as intolerance to oral feeds requiring nasogastric aspiration after the sixth postoperative day.
Wound Infection (Infections and infestations) | 4 (4) — Wound Infection was defined as purulent discharge from the main wound with positive culture report.
Intraabdominal Abscess (Infections and infestations) | 2 (2) — Intraabdominal Abscess was defined as purulent fluid of any amount inside the abdomen requiring percutaneous drainage or laparotomy.
Postoperative Fever (General disorders) | 2 (2) — Postoperative fever was defined as core body temperature more than 100 F sustained enough to require medication and search for its cause after surgery.

LIMITATIONS AND CAVEATS:
The analysis was done from a prospectively maintained database and target followup done for a period of 5 years after surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No